CLINICAL TRIAL: NCT02760550
Title: Policy-Related Survey - Territory-wide Telephone Survey on Tobacco Control
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Robert Kotewall Professor in Public Health, The University of Hong Kong
Other Study IDs: 2015 Policy Survey
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- never smokers: who have never smoked at all
  Interventions: Other: No intervention
- ex-smokers: formerly smokers but currently do not smoke at all
  Interventions: Other: No intervention
- current smokers: current smokers who, at the time of the survey, smoke any tobacco product either daily or occasionally. Social smokers fall into this category and are defined as those who smoke less than one cigarette per week or smoke only in some occasions
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants of all three groups completed a questionnaire.

SUMMARY:
The objectives of this policy-related survey are as follows:

i. to study updated trend and prevalence on secondhand smoke, smoking-attributed health effects, cessation services; ii. to investigate the level of public support on current and future tobacco control measures and taxation policies; iii. to address the timely impacts of smoke-free policies, substantiate public support on further tobacco control measures and assist Hong Kong Council On Smoking and Health (COSH) in shaping policy direction for government.

Purpose of the study is to provide evidence and support for smoke-free policy development in Hong Kong.

DETAILED DESCRIPTION:
Smoking is a major cause of premature death. Each year, tobacco kills nearly 6 million people globally, including more than 600,000 non-smokers by secondhand smoke (SHS). During the past few decades, tobacco control has contributed prominently to international health, and the World Health Organization (WHO) Framework Convention on Tobacco Control (FCTC), the first international health treaty negotiated by WHO has propelled tobacco control into a new era. In order to determine the impact of and opinions on tobacco control policies, many countries around the world have carried out surveys on policies either implemented or under consideration. A number of surveys have assessed the impact of policies such as smoke-free laws, including the National Health and Nutrition Examination Survey (NHANES), the International Tobacco Control (lTC) Surveys and the Global Adult Tobacco Survey (GATS).

In 2013 and 2014, the investigators conducted two waves of the policy-related survey on tobacco control. The surveys gathered information such as SHS exposure at home, in the workplace, and in various public places (e.g. bars/restaurants, door way of the buildings, streets, and bus stops), use of smoking cessation services, knowledge of smoking and quitting, and smoking prevalence; measured the impact of tobacco control policies such as tax increase in 2011 and 2014, expansion of smoke-free areas in 2009 and 2010, and pictorial health warnings on behavioural change of smokers and ex-smokers; collected the opinions on current policies such as smoke-free areas, pictorial health warnings and point of sale displays, and the opinions towards future policies such as tax increase, plain packaging, and tobacco endgame. The results of the two waves have been used by COSH to advocate plain packaging, banning on point of sale displays, and increasing tobacco tax by 100% in the past 2 years.

In order to collect further information on issues related to tobacco control which should be addressed in future tobacco control measures in Hong Kong, COSH commissioned School of Public Health (SPH), the University of Hong Kong (HKU), to conduct a third wave of the survey (2014/15). The current survey sought to use the Hong Kong data to update information on the prevalence of SHS and active smoking and its health effects, use of E-cigarettes, awareness of smoking cessation services and to identify the level of public support for current and future tobacco control measures as well as estimating the impact of existing policies.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese speakers

Exclusion Criteria:

* Unable to provide a consent form
* Speak language other than Cantonese

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hong Kong residents
Sampling Method: Probability Sample
Enrollment: 5252 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The prevalence of active smoking in Hong Kong | Outcome will be assessed immediately after subjects answer the questionnaire as this is a cross-sectional survey

SECONDARY OUTCOMES:
The prevalence of secondhand smoking in Hong Kong | Outcome will be assessed immediately after subjects answer the questionnaire as this is a cross-sectional survey
The prevalence of e-cigarette in Hong Kong | Outcome will be assessed immediately after subjects answer the questionnaire as this is a cross-sectional survey

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — School of Public Health, the University of Hong Kong

IPD SHARING:
Plan to Share IPD: No